CLINICAL TRIAL: NCT06400303
Title: KYSA-5: A Phase 1/2, Open-Label, Multicentre Study of KYV 101, an Autologous Fully Human Anti-CD19 Chimeric Antigen Receptor T Cell (CD19 CAR T) Therapy, in Subjects With Systemic Sclerosis
Brief Title: KYSA-5: A Study of Anti-CD19 Chimeric Antigen Receptor T-Cell (CD19 CAR T) Therapy, in Subjects With Systemic Sclerosis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kyverna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KYSA-5; KYV101-005 (Other: Kyverna Therapeutics)
Record Dates: First submitted 2023-08-29; First posted 2024-05-06 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Systemic Sclerosis; Systemic Sclerosis - Diffuse Cutaneous; Systemic Sclerosis - 2013 ACR/EULAR Classification Criteria
Keywords: KYV-101; systemic sclerosis; autoimmune disease; anti-CD19 CAR-T therapy; cellular therapy; Scleroderma
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Autoimmune Diseases | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KYV-101 CAR-T cells with lymphodepletion conditioning (Phase 1) (Experimental): Dosing with KYV-101 CAR T cells
  Interventions: Biological: KYV-101; Drug: Standard lymphodepletion regimen
- KYV-101 CAR-T cells with lymphodepletion conditioning (Phase 2) (Experimental): Recommended Phase 2 Dose
  Interventions: Biological: KYV-101; Drug: Standard lymphodepletion regimen

INTERVENTIONS:
Biological: KYV-101 — Anti-CD19 CAR-T cell therapy
Drug: Standard lymphodepletion regimen — Standard lymphodepletion regimen
  Other Names: Cyclophosphamide; Fludarabine

SUMMARY:
A Study of Anti-CD19 Chimeric Antigen Receptor T Cell Therapy for Subjects with Systemic Sclerosis

DETAILED DESCRIPTION:
SSc is an immune-mediated rheumatic disease that is characterized by fibrosis of the skin and internal organs and vasculopathy. B-cells play a role in SSc, and the disease is characterized by the presence of autoantibodies such as anti-Scl-70 and anti-RNAP III antibodies. CD19-targeted chimeric antigen receptor (CAR) T-cells harness the ability of cytotoxic T-cells to directly and specifically lyse target cells to effectively deplete B-cells in the circulation and in lymphoid and potentially non-lymphoid tissues. KYV-101, a fully human anti-CD19 CAR T-cell therapy, will be investigated in adult subjects with systemic sclerosis.

ELIGIBILITY:
Key Inclusion Criteria

1. Clinical diagnosis of SSc according to 2013 ACR/EULAR classification
2. Clinical disease as follows: Classified as diffuse cutaneous SSc; ≤ 6 years since first non-Raynaud's sign or symptom; active disease
3. Up to date on all recommended vaccinations per CDC or institutional guidelines for immune-compromised individuals

Key Exclusion Criteria

1. Clinically significant ILD
2. Prior treatment with cellular therapy (CAR-T) or gene therapy product directed at any target
3. History of allogeneic or autologous stem cell transplant
4. Evidence of active hepatitis B or hepatitis C infection
5. Positive serology for HIV
6. Primary immunodeficiency
7. History of splenectomy
8. History of stroke, seizure, dementia, Parkinson's disease, coordination movement disorder, cerebellar diseases, psychosis, paresis, aphasia, and any other neurologic disorder investigator considers would increase the risk for the subject
9. Impaired cardiac function or clinically significant cardiac disease
10. Previous or concurrent malignancy with the following exceptions:

    1. Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to screening)
    2. In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to screening
    3. A primary malignancy which has been completely resected, or treated, and is in complete remission for at least 5 years prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and laboratory abnormalities (Phase 1) | Up to 2 years
Frequency of Dose-Limiting Toxicities (DLTs) at each dose level (Phase 1) | Up to 2 years
To evaluate efficacy of KYV-101(Phase 2) | 52 weeks
  via revised Composite Response Index in Systemic Sclerosis (rCRISS) 30/5

SECONDARY OUTCOMES:
To evaluate pharmacodynamics (PK) of KYV-101 in blood (Phase 1 and Phase 2) | Up to 2 years
  Chimeric antigen receptor-positive (CAR-positive) T-cell counts in blood
To evaluate pharmacodynamics (PD) of KYV-101 in blood (Phase 1 and Phase 2) | Up to 2 years
  Levels of B-cells in blood
To evaluate pharmacodynamics (PD) of KYV-101 in blood (Phase 1 and Phase 2) | Up to 2 years
  Levels of cytokines in serum
To evaluate efficacy of KYV-101 (Phase 1 and Phase 2) | 12, 24, 52 weeks
  revised Composite Response Index in Systemic Sclerosis (rCRISS) 30/5 response rate
To evaluate immunogenicity (humoral response) of KYV-101 (Phase 1 and Phase 2) | Up to 2 years
  Percentage of participants who develop anti-KYV-101 antibodies by immunoassays
To define the Recommended Phase 2 Dose (RP2D) (Phase 1) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Kyverna Therapeutics, Inc.
Locations (2):
- United States (2):
  - Stanford University Medical Center, Palo Alto, California
  - Northwell Health, Great Neck, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bosello S, Angelucci C, Lama G, Alivernini S, Proietti G, Tolusso B, Sica G, Gremese E, Ferraccioli G. Characterization of inflammatory cell infiltrate of scleroderma skin: B cells and skin score progression. Arthritis Res Ther. 2018 Apr 18;20(1):75. doi: 10.1186/s13075-018-1569-0. PMID 29669578